CLINICAL TRIAL: NCT02483858
Title: Phase I Study of Oral PQR309 in Patients With Advanced Solid Tumors
Brief Title: Study of Oral PQR309 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PIQUR Therapeutics AG (Industry)
Collaborators: Roswell Park Cancer Institute (Other); M.D. Anderson Cancer Center (Other); Mayo Clinic (Other); Hospital Clinic of Barcelona (Other); University College London Hospitals (Other); Churchill Hospital (Other); Case Western Reserve University (Other); University Hospital, Zürich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PQR309-003
Record Dates: First submitted 2015-05-19; First posted 2015-06-29 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Cancer
Keywords: oncology, solid tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PQR309 (Experimental): Different dose Evaluation (continous and intermittent) 20-160mg daily
  Interventions: Drug: PQR 309

INTERVENTIONS:
Drug: PQR 309 — Intervention of this drug may include safety, tolerability, PK (pharmacokinetics) and efficacy
  Other Names: PI3K/mTOR/AKT Inhibitor

SUMMARY:
This is an open-label, multi-center, non-randomized, dose escalation Phase 1 study evaluating safety, tolerability, PK (pharmacokinetics) and efficacy of PQR309 in the treatment of selected patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is an open-label, multi-center, non-randomized, dose escalation Phase 1 study evaluating safety, tolerability, PK (pharmacokinetics)and efficacy of PQR309 in the treatment of selected patients with advanced solid tumors.

In the initial phase of the study, patients will be treated once daily until disease progression, unacceptable toxicity, patient's request for withdrawal, investigator judgment or death whichever comes first. Enrollment of an initial patient cohort of 3 or 6 patients will follow the traditional 3 + 3 dose escalation scheme to evaluate Dose Levels 1 - 5 with continuous q.d dosing schedule. Patients will be treated with PQR309 at starting Dose Level 1 enrolling exceptionally 6 patients (only applicable for continuous dosing schedule). Subsequent patient cohort(s) will be enrolled depending on the safety and tolerability of the initial cohort. If < 33% patients treated at Dose Level 1 (80 mg) experience Dose Limiting Toxicities (DLT - see definition below) by the end of first treatment cycle (21 days), next cohort of 3 patients will be enrolled and treated at Dose Level 2 of the continuous dosing schedule, if 2 or more treatment-related DLTs are observed at Dose Level 1, patients will be accrued to Dose Level -1. If 2 or more patients experience a DLT during dose Level 2 (120 mg), the dose of 100 mg will be explored next.The MTD is defined as the maximum dose level at which ≤ 1/6 patients have DLTs. After the MTD has been established with the continuous dosing schedule, the study will be expanded to evaluate the MTD of intermittent dosing schedules. Initially 2 additional dosing schedules, intermittent schedule A and B, will be evaluated in parallel. Patients will be assigned to the two schedules in an alternating manner.

Patients will be treated only within dose and schedule cohort they have been enrolled in. No within-patient dose escalation or alteration of dosing schedule will be allowed.Both schedules A and B will evaluate intermittent dosing in 21 day cycles:

Intermittent schedule A:

Two days of once daily PQR309 administration followed by no treatment for 5 days.

Intermittent schedule B:

PQR309 administration on Monday and Thursday. Same dose escalation procedures will apply to intermittent schedule evaluation as for the continuous schedule. Based on the overall evaluation of safety and tolerability, the PK (pharmacokinetics) data of the intermittent dosing schedules and the continuous schedule as well as PQR309 non-clinical data, evaluation of additional dosing schedules may be considered and investigated if agreed between sponsor and study investigators.

After the MTD has been established with the intermittent dosing schedules, the study will be expanded to evaluate the MTD of one selected schedule in patients with:

* Solid tumors with PI3K/mTOR pathway activation
* HPV positive HNSCC patients containing activating PIK3CA mutations Evaluation of the data from these cohorts will allow for more complete evaluation of tolerability, pharmacokinetics, and correlative endpoints as well as the preliminary clinical efficacy of PQR309.

ELIGIBILITY:
Inclusion Criteria

1. Patients ≥ 18 years of age.
2. Histologically or cytologically confirmed diagnosis of solid malignancy, for which no standard curative or life prolonging therapy is available.
3. Have an ECOG Performance Status of ≤ 1. Refer to Appendix 1.
4. Life expectancy of ≥ 12 weeks.
5. Adequate bone marrow, liver, and renal functions, defined as:

   * Platelet count ≥ 100 x 109/L, absolute neutrophil count (ANC)

     ≥ 1.5 x 109/L, Hemoglobin ≥ 9 g/dL.
   * ALT and AST ≤ 2.5 upper limit normal (ULN), or < 5 x ULN if liver metastases are present; serum total bilirubin ≤ ULN or 1.5 x ULN if liver metastases are present or total 3 x ULN with direct bilirubin ≤ ULN in patients with well documented Gilbert Syndrome.
   * Serum Creatinine < 1.5 x ULN (upper limit of normal) or estimated creatinine clearance ≥ 60 mL/min, as calculated using method standard for the institution (Appendix 2).
6. Glycated hemoglobin (HgbA1c) ≤ 7 %; Fasting Plasma Glucose (FPG) ≤ 7.0 mmol/L (125 mg/dL).
7. Women of childbearing potential must have a negative pregnancy test (urine or serum) performed within 7 days prior to the start of study drug.
8. Able and willing to swallow and retain oral medication.
9. Subject or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

   Expansion part:
10. Patients must have known PI3K/mTOR pathway gene aberrations (from molecular profiling studies).
11. Patients must have HPV positive HNSCC containing activating PIK3CA mutations.

Exclusion Criteria

1. Concurrent or previous anti-cancer chemotherapy, immunotherapy or investigational agents < 3 weeks, or palliative radiation < 2 weeks prior to the first day of study treatment. Patients who receive gamma knife radiosurgery for brain metastases or whole brain radiation are eligible if gamma knife radiosurgery was performed > 2 weeks before treatment is started or whole brain radiation was performed > 4 weeks before treatment is started, and are clinically stable.
2. Hormonal anticancer therapies except for LHRH antagonists or LHRH agonists in hormone-refractory prostate cancer
3. Patient has a known hypersensitivity to any of the excipients of PQR309.
4. Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects.
5. Patients with poorly controlled diabetes mellitus, steroid-induced diabetes mellitus, HbA1c > 7%, or FPG > 7.0 mmol/L (125 mg/dL).
6. Patients who are on (or will require) prolonged systemic corticosteroid treatment during the study, except for:

   * if receiving corticosteroids, patients must have been on a stable or decreasing dose of corticosteroids and no more than 1 mg of dexamethasone a day or equivalent, i.e. 6 mg prednisone or 25 mg hydrocortisone for at least 5 days prior to date of enrollment.
   * a short duration (< 5 days) of systemic corticosteroids e.g., of chronic obstructive pulmonary disease, or as an antiemetic corresponding at maximum to the anti-inflammatory potency of 4 mg dexamethasone for treatment;
   * topical applications for treatment of e.g., rash, inhaled sprays for treatment of e.g., obstructive airways diseases, eye drops or local Protocol No. PQR309-003 Protocol Amendment 3, 23 September 2015 PIQUR Therapeutics AG - Confidential Page 15 of 108 injections (e.g., intra-articular);
7. Patients who have taken herbal medications and certain fruits within 7 days prior to starting study drug, see section 11.1.2.7.
8. Patients who have other concurrent severe and/or uncontrolled medical conditions that would, in the investigator's judgment, contraindicate patient participation in the clinical study (e.g., active or uncontrolled severe infection, chronic active hepatitis, immuno-compromised, acute or chronic pancreatitis, uncontrolled high blood pressure, interstitial lung disease, etc.).
9. Patient has a known history of HIV infection (testing not mandatory).
10. Patient has any of the following cardiac abnormalities:

    * History of, or current, documented congestive heart failure (New York Heart Association functional classification III - IV), documented cardiomyopathy.
    * Left Ventricular Ejection Fraction (LVEF) < 40% as determined by Multiple Gated Acquisition (MUGA) scan or echocardiogram (ECHO).
    * Myocardial infarction ≤ 6 months prior to enrolment.
    * Unstable angina pectoris.
    * Serious uncontrolled cardiac arrhythmia.
    * Symptomatic pericarditis.
11. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug.
12. Concomitant treatment with medicinal products that increase the pH (reduce acidity) of the upper gastrointestinal tract, including, but not limited to, proton-pump inhibitors (e.g. omeprazole), H2-antagonists (e.g. ranitidine) and antacids. Patients may be enrolled in the study after a wash-out period sufficient to terminate their effect.
13. Patient has a history of non-compliance to medical regimen or inability to grant consent.
14. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive Human Chorionic Gonadotropin (hCG) laboratory test (> 5 mIU/mL). Patients with elevated hCG at baseline that is judged to be related to the tumor are eligible if hCG levels do not show the expected doubling when repeated 5 - 7 days later, or pregnancy has been ruled out by vaginal ultrasound.
15. Patient who does not apply highly effective contraception during the study from screening until 90 days after discontinuing study treatment Protocol No. PQR309-003 Protocol Amendment 3, 23 September 2015 PIQUR Therapeutics AG - Confidential Page 16 of 108 (see section 11.3).
16. Patients have any of the following mood disorders as judged by the Investigator or a Psychiatrist, or who meets the cut-off score of ≥ 12 the PHQ-9 or a cut-off of ≥ 15 in the GAD-7 mood scale, respectively, or selects a positive response of '1, 2, or 3' to question number 9 regarding potential for suicidal thoughts in the PHQ-9 (independent of the total score of the PHQ-9) see Appendix 4.

    * Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others).
    * ≥ CTCAE Grade 3 anxiety.
17. Patients with a history of interstitial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
To identify the Maximum Tolerated Dose (MTD) of PQR309 administered in different (continuous and intermittent) dosing schedules. To evaluate efficacy of PQR309 in selected patient population: • Solid tumors with PI3K/mTOR activation • Human Papilloma | In average 1 year
  MTD based on the rate of dose-limiting toxicities. The MTD is defined as the maximum dose level at which ≤ 1/6 patients have dose limiting toxicities (DLTs).
Objective response rate (ORR) according to the response evaluation• Solid tumors with PI3K/mTOR activation • Human Papilloma Virus (HPV) positive Head and neck squamous cell carcinoma (HNSCC) containing activating PIK3CA mutations | in average 2 years
  Expansion part criteria in solid tumors (RECIST), version 1.1

SECONDARY OUTCOMES:
Number of patients with adverse Events and serious adverse events | Cycle1 on Day1,8,15, Cycle 2 and subsequent cycles on Day 1, End of the treatment up to 3 days and as follow up 30 days after last dosing
  Continous Dosing and intermittent dosing "2days on/5days off
Number of patients with adverse Events and serious adverse events | Assessment on Day 1 after basline, Cycle1 on Day 8,15, Cycle 2 and subsequent cycles on Day 1, End of the treatment up to 3 days and as follow up 30 days after last dosing
  "Monday/ Thursday"
Physical examination according to ECOG (Eastern Cooperative Oncology Group) Performance Status | Cycle 1 on Day 8,15, Cycle 2 and subsequent cycles on Day1 , end of treatment up to 3 days after
  Continous Dosing
Physical examination according to ECOG (Eastern Cooperative Oncology Group) Performance Status | Cycle 1 on Day 1,8,15, Cycle 2 and subsequent cycles on Day1 , end of treatment up to 3 days after
  Intermittent Dosing "2days on/5days off"
Physical examination according to ECOG (Eastern Cooperative Oncology Group) Performance Status | Assessment on Day1,2, Cycle 1 on Day 4,8,9,15
  Intermittent Dosing "Monday/ Thursday"
Change in Pulse Rate | Assessment on Day 3 after baseline, Cycle 1 on Day 1,8,15, Cycle 2 and subsequent cycles on Day1, end of treatment up to 3 days after last medication
  Continous Dosing
Change in Pulse Rate | Cycle 1 on Day 1,8,15, Cycle 2 and subsequent cycles on Day1, end of treatment up to 3 days after last medication
  Intermittent Dosing "2 days on/5days off"
Change in Pulse Rate | Assessment on Day1,2,Cycle 1 on Day 4,8,9,15
  Intermittent Dosing "Monday/ Thursday"
Change in Temperature | Assessment on Day 3 after baseline, Cycle 1 on Day 1,8,15, Cycle 2 and subsequent cycles on Day1, end of treatment up to 3 days after last medication
  Continous Dosing
Change in Temperature | Cycle 1 on Day 1,8,15, Cycle 2 and subsequent cycles on Day1, end of treatment up to 3 days after last medication
  Intermittent Dosing "2days on/5days off"
Change in Temperature | Assessment on Day1,2,Cycle 1 on Day 4,8,9,15
  Intermittent Dosing " Assessment on Day1,2,Cycle 1 on Day 4,8,9,15
Change in Respiratory Rate | Assessment on Day 3 after baseline, Cycle 1 on Day 1,8,15, Cycle 2 and subsequent cycles on Day1, end of treatment up to 3 days after last medication
  Continous Dosing
Change in Respiratory Rate | Cycle 1 on Day 1,8,15, Cycle 2 and subsequent cycles on Day1, end of treatment up to 3 days after last medication
  Intermittent Dosing "2days on/5days off"
Change in Respiratory Rate | Assessment on Day1,2,Cycle 1 on Day 4,8,9,15
  Intermittent Dosing " Monday/ Thursday"
Change in Blood Pressure | Assessment on Day 3 after baseline, Cycle 1 on Day 1,8,15, Cycle 2 and subsequent cycles on Day1, end of treatment up to 3 days after last medication
  Continous Dosing
Change in Blood Pressure | Cycle 1 on Day 1,8,15, Cycle 2 and subsequent cycles on Day1, end of treatment up to 3 days after last medication
  Intermittent Dosing "2days on/5days off"
Change in Blood Pressure | Assessment on Day1,2,Cycle 1 on Day 4,8,9,15
  Intermittent Dosing "Monday/ Thursday"
Change in Blood Body Weight | Assessment on Day 3 after baseline, Cycle 1 on Day 1,8,15, Cycle 2 and subsequent cycles on Day1, end of treatment up to 3 days after last medication
  Continous Dosing
Change in Blood Body Weight | Cycle 1 on Day 1,8,15, Cycle 2 and subsequent cycles on Day1, end of treatment up to 3 days after last medication
  Intermittent Dosing "2days on/5days off"
Change in Blood Body Weight | Assessment on Day1,2,Cycle 1 on Day 4,8,9,15
  Intermittent Dosing "Monday/ Thursday"
Change in ECG | Assessment on Day 3 after baseline, Cycle 1 on Day 8,15, Cycle 2 and subsequent cycles on Day1, end of treatment up to 3 days after last medication
  Continous Dosing
Change in ECG | After Cycle 2 and subsequent cycles on Day1, end of treatment up to 3 days after last medication
  Intermittent Dosing "2days on/5days off" and "Monday/ Thursday"
Depression test (PHQ-9) | After Cycle 2 and subsequent cycles on Day1, end of treatment up to 3 days after last medication
  Continous Dosing
Depression test (PHQ-9) | Cycle 1 on Day 8,15, Cycle 2 and subsequent cycles on Day1, end of treatment up to 3 days after last medication
  Intermittent Dosing "2days on/5days off" and "Monday/ Thursday"
Generalized anxiety disorder mood scale score (GAD7) | Cycle 1 on Day 8,15, Cycle 2 and subsequent cycles on Day1, end of treatment up to 3 days after last medication
  Continous Dosing and Intermittent Dosing "2days on/5days off" and "Monday/ Thursday"
Changes in routine blood chemistry | Cycle 1 on Day 1, 8,15, Cycle 2 and subsequent cycles on Day1, end of treatment up to 3 days after last medication
  Continous Dosing and Intermittent Dosing "2days on/5days off"
Changes in routine blood chemistry | Assessment on Day 1 after baseline, Cycle 1 on Day 8,15, Cycle 2 and subsequent cycles on Day1, end of treatment up to 3 days after last medication
  Intermittent Dosing "Monday/ Thursday"
Changes of hematology | Cycle 1 on Day 1, 8,15, Cycle 2 and subsequent cycles on Day1, end of treatment up to 3 days after last medication
  Continous Dosing and Intermittent Dosing "2days on/5days off"
Changes of hematology | Assessment on Day 1 after baseline, Cycle 1 on Day 8,15, Cycle 2 and subsequent cycles on Day1, end of treatment up to 3 days after last medication
  Intermittent Dosing "Monday/ Thursday"
Changes of insulin/Glucose/ C-peptide | Assessment on Day 3, ,2,1 after baseline, Cycle 1 on Day 1, Cycle 2 and subsequent cycles on Day1
  Continous Dosing
Changes of insulin/Glucose/ C-peptide | Assessment on Day 3, 2,1 after baseline, Cycle 8,9,15 on Day 1
  " Intermittent Dosing "2days on/5days off""
Changes of insulin/Glucose/ C-peptide | Assessment on Day 1,2 after baseline, Cycle1 on Day 4, 8,9,15
  " Intermittent Dosing "Monday/ Thursday"
Changes of haemostasis | Cycle 1 on Day 1, 8, 15 Cycle 2 and subsequent cycles on Day1, end of treatment up to 3 days after last medication
  Continous Dosing and Intermittent Dosing "2days on/5days off"
Changes of haemostasis | Assessment on Day 1 after baseline, Cycle 1 on Day 1,15 Cycle 2 and subsequent cycles on Day1, end of treatment up to 3 days after last medication
  Intermittent Dosing "Monday/ Thursday"
Determination of Cmax | Assessment on Day 3,2,1 after baseline, Cycle 1 on Day 8,15, Cycle 2 on Day1
  Continous Dosing
Determination of Cmax | Assessment on Day 3,2,1 after baseline, Cycle 1 on Day 8,9,15
  Intermittent Dosing "2days on/5days off"
Determination of Cmax | Assessment on Day 1,2 after baseline, Cycle 1 on Day 4,8,9,15
  Intermittent Dosing "Monday/ Thursday"
Determination of AUC 0-24 | Assessment on Day 3,2,1 after baseline, Cycle 1 on Day 8,15, Cycle 2 on Day1
  Continous Dosing
Determination of AUC 0-24 | Assessment on Day 3,2,1 after baseline, Cycle 1 on Day 8,9,15
  Intermittent Dosing "2days on/5days off"
Determination of AUC 0-24 | Assessment on Day 1,2 after baseline, Cycle 1 on Day 4,8,9,15
  Intermittent Dosing "Monday/ Thursday"
Determination of tmax | Assessment on Day 3,2,1 after baseline, Cycle 1 on Day 8,15, Cycle 2 on Day1
  Continous Dosing
Determination of tmax | Assessment on Day 3,2,1 after baseline, Cycle 1 on Day 8,9,15
  Intermittent Dosing "2days on/5days off"
Determination of tmax | Assessment on Day 1,2 after baseline, Cycle 1 on Day 4,8,9,15
  Intermittent Dosing "Monday/ Thursday"
Determination of AUClast (area under the curve) | Assessment on Day 3,2,1 after baseline, Cycle 1 on Day 8,15, Cycle 2 on Day1
  Continous Dosing
Determination of AUClast | Assessment on Day 3,2,1 after baseline, Cycle 1 on Day 8,9,15
  Intermittent Dosing "2days on/5days off"
Determination of AUClast | Assessment on Day 1,2 after baseline, Cycle 1 on Day 4,8,9,15
  Intermittent Dosing "Monday/ Thursday"
Determination of AUC0-∞ | Assessment on Day 3,2,1 after baseline, Cycle 1 on Day 8,15, Cycle 2 on Day1
  Continous Dosing
Determination of AUC0-∞ | Assessment on Day 3,2,1 after baseline, Cycle 1 on Day 8,9,15
  Intermittent Dosing "2days on/5days off"
Determination of AUC0-∞ | Assessment on Day 1,2 after baseline, Cycle 1 on Day 4,8,9,15
  Intermittent Dosing "Monday/ Thursday"
Determination of t 1/2 | Assessment on Day 3,2,1 after baseline, Cycle 1 on Day 8,15, Cycle 2 on Day1
  Continous Dosing
Determination of t 1/2 | Assessment on Day 3,2,1 after baseline, Cycle 1 on Day 8,9,15
  Intermittent Dosing "2days on/5days off"
Determination of t 1/2 | Assessment on Day 1,2 after baseline, Cycle 1 on Day 4,8,9,15
  Intermittent Dosing "Monday/ Thursday"
Determination of RAC (Accumulation Ratio) | Assessment on Day 3,2,1 after baseline, Cycle 1 on Day 8,15, Cycle 2 on Day1
  Continous Dosing
Determination of RAC (Accumulation Ratio) | Assessment on Day 3,2,1 after baseline, Cycle 1 on Day 8,9,15
  Intermittent Dosing "Monday/ Thursday"
Determination of RAC (Accumulation Ratio) | Assessment on Day 1,2 after baseline, Cycle 1 on Day 4,8,9,15
  Intermittent Dosing "Monday/ Thursday"
Determine Time to Response (TTR) | up to 2 years
  Efficacy
Determine Duration of Response (DOR) | baseline and on Day 1 of every subsequential cycle which can be up to 24 months
  Defined as the time from the date of the first confirmed response to the first documentation of relapse or progressive disease, whichever occurs first
Time to Treatment Failure (TTF) | Tumor Measurement preferably with a ruler and/or MRI scans e.g. and incorporated clinical signs will be assesses at baseline and on Day 1 of every subsequential cycle which can be up to 24 months
  Defined as the time from study entry to any treatment failure including disease progression or discontinuation of treatment for any reason (e.g., disease progression, AE, patient preference, initiation of new treatment without documented progression, death)
Determine Progression Free Survival (PFS) | baseline and on Day 1 of every subsequential cycle which can be up to 24 months
  Defined as the time from study entry to progression or death due to any cause
1- year Survival Rate | baseline and on Day 1 of every subsequential cycle which can be up to 36 months
  Defined as the time from study entry to death as a result of any cause at 1-year cutoff date

CONTACTS AND LOCATIONS:
Overall Officials: Mateusz Opyrchal, Study Director — Roswell Park Cancer Institute; Filip Janku, Principal Investigator — MD Anderson Cancer; Afshin Dowlati, Principal Investigator — University Hospitals Cleveland Medical Center; Alex Adjei, Principal Investigator — Mayo Clinic; Jordi Rodon, Principal Investigator — Vall d'Hebron University Hospital; Martin Forster, Principal Investigator — University College London Hospitals; Sarah Bladgen, Principal Investigator — Chruchill Hospital; Andreas Wicki, Principal Investigator — Basel University Hospital
Locations (1):
- M.D. Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided